CLINICAL TRIAL: NCT01274676
Title: Randomized Trial of Proximal-versus Distal Cerebral Protection on Micro Embolization During Carotid Artery Stenting in Patients With High Risk Lipid Palque
Brief Title: Carotid Stenting in Patients With High Risk Carotid Stenosis ("Soft Plaque")
Acronym: MOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Piero Montorsi, MD, Centro Cardiologico Monzino, IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S111/508
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2009-09

CONDITIONS: Carotid Stenosis
Keywords: stenting; carotid plaque; stenosis; angioplasty
MeSH Terms: conditions — Carotid Stenosis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carotid stenting with MOMA (Active Comparator)
  Interventions: Device: carotid stenting with MOMA
- Carotid stenting with filter wire EZ (Active Comparator)
  Interventions: Device: Carotid stenting with filter wire EZ

INTERVENTIONS:
Device: carotid stenting with MOMA — The MOMA system is an endovascular catheter for proximal protection during carotid stenting. The system allows a concomitant balloon occlusion of both external and common carotid arteries leading to blood flow reversal within the internal carotid artery.
  Other Names: MOMA device (INVATEC RONCADELLE, BRESCIA - ITALY)
  Arms: carotid stenting with MOMA
Device: Carotid stenting with filter wire EZ — The filter wire EZ a distal protection system that is placed in he distal internal carotid artery before carotid stenting. The filter should entrap almost all the debries that are generated during endovascular procedure. At the end of the procedure the filter is retrieved throught a dedicated retrieval catheter.
  Other Names: Filterwire EZ - Boston Scientific
  Arms: Carotid stenting with filter wire EZ

SUMMARY:
Stenting is an alternative to traditional surgery in the treatment of carotid stenosis.The intra and/or postprocedural cerebral embolization remains the most frequent complication. Thanks to the systematic use of cerebral protection systems, these complications have reduced.A debate concerning which cerebral protective device should be more effective is still ongoing.

ELIGIBILITY:
Inclusion Criteria:

-patients with monolateral, significant, soft carotid stenosis

Exclusion Criteria:

* patients with controlateral carotid occlusion
* patients with critic stenosis of the external carotid

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
number of Microembolization signals (MES) detected with transcranal doppler | 6 different phases of carotid stenting (lesion wiring; predilation; stent crossing of the lesion; stent deployment; stent post dilation; device tetruieval/deflation

SECONDARY OUTCOMES:
Clinical success | In hospital and 30 days
  Assesment of any clinical and neurological complication (death, any stroke, TIA; myocardial infarction).

CONTACTS AND LOCATIONS:
Overall Officials: Piero Montorsi, MD, Principal Investigator — Centro Cardiologico Monzino, IRCCS
Locations (1):
- Centro Cardiologico Monzino, IRCCS, Milan, Italy

REFERENCES:
- [Derived] Montorsi P, Caputi L, Galli S, Ciceri E, Ballerini G, Agrifoglio M, Ravagnani P, Trabattoni D, Pontone G, Fabbiocchi F, Loaldi A, Parati E, Andreini D, Veglia F, Bartorelli AL. Microembolization during carotid artery stenting in patients with high-risk, lipid-rich plaque. A randomized trial of proximal versus distal cerebral protection. J Am Coll Cardiol. 2011 Oct 11;58(16):1656-63. doi: 10.1016/j.jacc.2011.07.015. PMID 21982309